CLINICAL TRIAL: NCT00422006
Title: Study of the Role of PCSK9 and FXR in the Physiopathology of the Joint Dyslipidemia Associated to the Human Immunoresistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BRD 06/8-I; ID RCB 2006-A00196-45; DGS2006-0090
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Obesity
Keywords: bariatric surgery planned
MeSH Terms: conditions — Obesity | interventions — Liver Extracts; Diet; Biopsy; Biological Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Non diabetic non dyslipidemic patient
  Interventions: Procedure: biopsy of muscle, of liver, and of adipose tissue; Procedure: clamp euglycemic - hyperglycemic; Behavioral: diet; Other: biopsies for biological and genetic analyses
- 2 (Experimental): Patient with metabolic syndrome
  Interventions: Procedure: biopsy of muscle, of liver, and of adipose tissue; Procedure: clamp euglycemic - hyperglycemic; Behavioral: diet; Other: biopsies for biological and genetic analyses
- 3 (Experimental): Patients with type II diabetes
  Interventions: Procedure: biopsy of muscle, of liver, and of adipose tissue; Procedure: clamp euglycemic - hyperglycemic; Behavioral: diet; Other: biopsies for biological and genetic analyses
- 4 (Experimental): Patient with a single lipidic anomaly
  Interventions: Procedure: biopsy of muscle, of liver, and of adipose tissue; Procedure: clamp euglycemic - hyperglycemic; Behavioral: diet; Other: biopsies for biological and genetic analyses

INTERVENTIONS:
Procedure: biopsy of muscle, of liver, and of adipose tissue — biopsy of muscle, of liver, and of adipose tissue
Procedure: clamp euglycemic - hyperglycemic — clamp euglycemic-hyperglycemic
Behavioral: diet — diet
Other: biopsies for biological and genetic analyses — biopsies for biological and genetic analyses

SUMMARY:
Experimental results are strongly suggesting that PCSK9 and FXR could occur in the physiopathology of human joined dyslipidemia. But no data in the literature can validate the potential role of these two genes in the lipidic and glucidic metabolism control in physiopathological situations. This protocol is based on the hypothesis that the expression levels of PCSK 9 and FXR are modified for some patients suffering from insulin resistance and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* corporal mass index > 40 kg/m² or > 35 kg/m² associated to a co-morbidity resistant to a diet
* bariatric surgery planned
* no lipid-lowering drugs during 4 weeks before surgery
* no treatment by metformin during 4 weeks before surgery
* no treatment by glitazones during 8 weeks before surgery
* age of the patient between 18 and 65 years
* consent form signed
* patient with social insurance

Exclusion Criteria:

* age inferior to 18 years
* women pregnant
* coagulation troubles
* surgery contraindicated
* Chronic hepatitis B or C active
* VIH infected
* other chronic hepatic disease
* patient with dyslipidemia under lipid-lowering drugs in secondary prevention of a cardiovascular pathology
* Type 2 diabetes under insulinosensitivator treatments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the relationship between the expression levels of PCSK9 and FXR in the liver, adipose tissue and muscle and the different components of the insulin resistance syndrome obese patients submitted to bariatric surgery | 2 years

SECONDARY OUTCOMES:
Relationship between the levels of hepatic expression of PCSK9 and FXR and the degree of NASH in these patients. - Search for mutations and polymorphisms in the gene PCSK9 and FXR and their promoter regions | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Cariou, MD, Principal Investigator — Nantes University Hospital; Michel Krempf, MD, Principal Investigator — Nantes University Hospital; Yassine Zaïr, MD, Principal Investigator — Nantes University Hospital; Eric Letessier, MD, Principal Investigator — Nantes University Hospital; Charles Couet, MD, Principal Investigator — CHU de Tours; Noël Huten, MD, Principal Investigator — CHU de Tours; Philippe Topart, MD, Principal Investigator — CHU de Brest; David Lechaux, MD, Principal Investigator — CHU de St Brieuc; Jean-Pierre Faure, MD, Principal Investigator — Poitiers University Hospital
Locations (1):
- CHU de Nantes, Nantes, France

REFERENCES:
- [Derived] Blanchard C, Ledoux S, Verhaegen A, Wargny M, Letessier E, Stepanian A, Huten N, Jacobi D, Krempf M, Le Bras M, Perrocheau Guillouche M, Arnaud L, Pichelin M, Van Gaal L, Cariou B, Le May C. Roux-en-Y gastric bypass, but not sleeve gastrectomy, decreases plasma PCSK9 levels in morbidly obese patients. Diabetes Metab. 2020 Nov;46(6):480-487. doi: 10.1016/j.diabet.2020.01.003. Epub 2020 Feb 4. PMID 32032671